CLINICAL TRIAL: NCT00973141
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-42160443 as Adjunctive Therapy in Subjects With Moderate to Severe Knee or Hip Pain From Osteoarthritis
Brief Title: A Dose-ranging Study of the Safety and Effectiveness of JNJ-42160443 as add-on Treatment in Patients With Osteoarthritis-related Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistic reasons associated with the FDA-imposed clinical hold.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016471; 42160443PAI2004 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.); 2009-009856-19 (EudraCT Number)
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee; Pain; Arthralgia; Joint Pain
Keywords: Moderate to severe, osteoarthritis-related pain; Osteoarthritis-related pain; Moderate to severe chronic pain; JNJ-42160443
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Osteoarthritis, Knee; Pain; Arthralgia | interventions — fulranumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (6):
- JNJ-42160443 1mg every 4 weeks (Experimental)
  Interventions: Drug: JNJ-42160443
- JNJ-42160443 3mg every 4 weeks (Experimental)
  Interventions: Drug: JNJ-42160443
- JNJ-42160443 3mg every 8 weeks (Experimental)
  Interventions: Drug: JNJ-42160443
- JNJ-42160443 6mg every 8 weeks (Experimental)
  Interventions: Drug: JNJ-42160443
- JNJ-42160443 10mg every 8 weeks (Experimental)
  Interventions: Drug: JNJ-42160443
- Matching placebo every 4 or 8 weeks (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42160443 — Type=exact number, unit=mg, number=1, form=solution for injection, route=Subcutaneous use. One injection of 1 mg of JNJ-42160443 every 4 weeks for up to 104 weeks (JNJ-42160443 at a concentration of 10 mg/mL was provided for use in this study).
  Arms: JNJ-42160443 1mg every 4 weeks
Drug: JNJ-42160443 — Type=exact number, unit=mg, number=10, form=solution for injection, route=Subcutaneous use. One injection of 10 mg of JNJ-42160443 every 8 weeks for up to 104 weeks (JNJ-42160443 at a concentration of 10 mg/mL was provided for use in this study).
  Arms: JNJ-42160443 10mg every 8 weeks
Drug: JNJ-42160443 — Type=exact number, unit=mg, number=3, form=solution for injection, route=Subcutaneous use. One injection of 3 mg of JNJ-42160443 every 8 weeks for up to 104 weeks (JNJ-42160443 at a concentration of 10 mg/mL was provided for use in this study).
  Arms: JNJ-42160443 3mg every 8 weeks
Drug: Placebo — Form=solution for injection, route=Subcutaneous injection. One injection of matching placebo every 4 or 8 weeks for up to 104 weeks.
  Arms: Matching placebo every 4 or 8 weeks
Drug: JNJ-42160443 — Type=exact number, unit=mg, number=3, form=solution for injection, route=Subcutaneous use. One injection of 3 mg of JNJ-42160443 every 4 weeks for up to 104 weeks (JNJ-42160443 at a concentration of 10 mg/mL was provided for use in this study).
  Arms: JNJ-42160443 3mg every 4 weeks
Drug: JNJ-42160443 — Type=exact number, unit=mg, number=6, form=solution for injection, route=Subcutaneous use. One injection of 6 mg of JNJ-42160443 every 8 weeks for up to 104 weeks (JNJ-42160443 at a concentration of 10 mg/mL was provided for use in this study).
  Arms: JNJ-42160443 6mg every 8 weeks

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of different doses of JNJ-42160443 with placebo in the treatment of chronic, moderate to severe knee or hip pain in patients with a diagnosis of osteoarthritis.

DETAILED DESCRIPTION:
This current study is a randomized (study drug assigned by chance), double-blind (neither the physician nor the patient knows the name of the assigned drug) study to evaluate the safety and effectiveness of different doses of JNJ-42160443 compared with placebo in the treatment of patients with a diagnosis of osteoarthritis of the hip or the knee who have moderate to severe pain that is not controlled by standard pain medications.Osteoarthritis is a chronic disease that affects the joints, and is characterized by degeneration of cartilage and bone. The duration of the study is approximately 133 weeks (3-week screening phase, 12-week double-blind efficacy phase, 92-week double-blind extension phase, and 26-week post treatment phase).JNJ-42160443 (10 mg/mL) or matching placebo given as an subcutaneous (injection under the skin) (SC) once every 4 weeks will be administered in the study as 1 of 5 JNJ-42160443 dosages:1 mg every 4 weeks, 3 mg every 4 weeks, 3 mg every 8 weeks, 6 mg every 8 weeks; or 10 mg every 8 weeks, or matching placebo for up to approximately 104 weeks (12-week double-blind efficacy phase + 92-week double-blind extension phase).

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of osteoarthritis of the hip or the knee; Have an average daily pain intensity score of >=5 averaged over the last 3 days before treatment assignment; Receiving a stable dose of non-steroidal anti-inflammatory drugs for a minimum of 5 days each week for the 4 weeks before screening or a stable dose of immediate-release opioids for a minimum of 5 days each week for the 4 weeks before screening, but not exceeding 200 mg oral morphine equivalents per day or a stable dose of long acting opioids for the 4 weeks before screening; but not exceeding 200 mg oral morphine equivalents per day; Have a mini mental state examination score of >=26 at screening. Exclusion Criteria:History within the past year of any of the following: seizure disorder; intrathecal therapy and ventricular shunts, mild or moderate traumatic brain injury, stroke, transient ischemic attack, meningitis; History of brain injury within the past 15 years consisting of >= 1 of the following, or with residual sequalae suggesting transient changes in consciousness: brain contusion, intracranial hematoma, either unconsciousness or posttraumatic amnesia lasting more than 24 hours; History of epilepsy or multiple sclerosis; Current diagnosis of fibromyalgia, complex regional pain syndrome (including reflex sympathetic dystrophy or causalgia), study joint pain caused by secondary infection, or pain caused by confirmed or suspected neoplasm; Any new or unresolved neurologic deficits, including progressive deficits, within 6 months before screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2009-09-16 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the average osteoarthritis-related pain intensity score | At the end of the 12-week double-blind efficacy phase

SECONDARY OUTCOMES:
Change from baseline in average OA-related pain intensity scores | At Weeks 4 and 8 and over the entire double-blind efficacy phase
Change from baseline in Pain, stiffness, and function subscales of the WOMAC 3.1 | At the end of the 12-week double-blind efficacy phase
Change from baseline in Pain severity and pain interference subscales of the BPI SF | At the end of the 12-week double-blind efficacy phase
Changes in PGA scores | At the end of the 12-week double-blind efficacy phase

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (77):
- United States (52):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carmichael, California
  - Fresno, California
  - Garden Grove, California
  - Pismo Beach, California
  - Roseville, California
  - San Diego, California
  - Clearwater, Florida
  - Jacksonville, Florida
  - Oldsmar, Florida
  - Port Orange, Florida
  - Tampa, Florida
  - Woodstock, Georgia
  - Boise, Idaho
  - Meridian, Idaho
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Valparaiso, Indiana
  - West Des Moines, Iowa
  - Prairie Village, Kansas
  - Topeka, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Lake Charles, Louisiana
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Rockville, Maryland
  - Hyannis, Massachusetts
  - Watertown, Massachusetts
  - East Lansing, Michigan
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - New York, New York
  - Williamsville, New York
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Duncansville, Pennsylvania
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Roanoke, Virginia
  - Spokane, Washington
- Canada (16):
  - Burnaby, British Columbia
  - Kamloops, British Columbia
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - St. John's, Newfoundland and Labrador
  - Brampton, Ontario
  - Cambridge, Ontario
  - Greater Sudbury, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Newmarket, Ontario
  - Sarnia, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- Poland (6):
  - Bialystok
  - Elblag
  - Gdynia
  - Lublin
  - Torun
  - Warsaw
- South Korea (3):
  - Busan
  - Daegu
  - Gwangju

REFERENCES:
- [Derived] Sanga P, Katz N, Polverejan E, Wang S, Kelly KM, Haeussler J, Thipphawong J. Long-Term Safety and Efficacy of Fulranumab in Patients With Moderate-to-Severe Osteoarthritis Pain: A Phase II Randomized, Double-Blind, Placebo-Controlled Extension Study. Arthritis Rheumatol. 2017 Apr;69(4):763-773. doi: 10.1002/art.39943. Epub 2017 Mar 8. PMID 27748055